CLINICAL TRIAL: NCT04012008
Title: Standard Versus Comprehensive Care for Post Acute Kidney Injury: A Randomized Controlled Trial
Brief Title: Standard Versus Comprehensive Care for Post Acute Kidney Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chulalongkorn University (Other)
Responsible Party: Principal Investigator, Nattachai Srisawat ,M.D., Associate Professor, Chulalongkorn University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Health Services Research
Other Study IDs: IRB.005/62
Record Dates: First submitted 2019-07-04; First posted 2019-07-09 (Actual); Last update posted 2022-10-31 (Actual); Status verified 2022-10

CONDITIONS: Acute Kidney Injury
MeSH Terms: conditions — Acute Kidney Injury | interventions — Comprehensive Health Care; Standard of Care

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard care (Active Comparator): * Regular follow-up by internists every 3 month
  * May consult nephrologists case-by-case
  Interventions: Other: Standard care
- Comprehensive care (Experimental): * Regular follow-up by nephrologists every 1-3 month
  * Multidisciplinary team consisting pharmacists, nurses, and dieticians
  Interventions: Other: Comprehensive care

INTERVENTIONS:
Other: Comprehensive care — * Regular follow-up by nephrologists every 1-3 month
  * Multidisciplinary team consisting pharmacists, nurses, and dieticians
  Arms: Comprehensive care
Other: Standard care — * Regular follow-up by internists every 3 month
  * May consult nephrologists case-by-case
  Arms: Standard care

SUMMARY:
The investigators aim to compare between standard versus comprehensive care for post-acute kidney injury who are admitted with acute kidney injury at least stage 2 or receive renal replacement therapy.

ELIGIBILITY:
Inclusion Criteria:

* Acute kidney injury at least stage 2 OR
* Received renal replacement therapy

Exclusion Criteria:

* Post kidney transplantation
* End-stage renal disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2019-07-16 (Actual); Primary Completion 2022-07-16 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
1 year major adverse kidney events | 1-year

CONTACTS AND LOCATIONS:
Locations (1):
- Chulalongkorn University, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Thanapongsatorn P, Chaikomon K, Lumlertgul N, Yimsangyad K, Leewongworasingh A, Kulvichit W, Sirivongrangson P, Peerapornratana S, Chaijamorn W, Avihingsanon Y, Srisawat N. Comprehensive versus standard care in post-severe acute kidney injury survivors, a randomized controlled trial. Crit Care. 2021 Aug 31;25(1):322. doi: 10.1186/s13054-021-03747-7. PMID 34465357